CLINICAL TRIAL: NCT00951977
Title: Live Kidney Donor Study - Cross-Sectional and Historical Cohort Study
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: DAIT RELIVE-04
Record Dates: First submitted 2009-07-31; First posted 2009-08-04 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: End Stage Renal Disease; Transplantation
Keywords: End Stage Renal Disease (ESRD); Transplantation; Living Kidney Donation; Kidney Transplant
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Subjects who have formerly donated a kidney
- Matched community control Subjects

SUMMARY:
Kidney transplantation from living donors has been shown to carry many benefits over deceased donor transplantation. Because of benefits such as shorter waiting times and improved outcome for transplant recipients, living kidney donation accounts for an increasing number of kidney transplants nationwide. Most published studies about living kidney donation demonstrate that the procedure is safe, but they also emphasize concerns that long-term data on live donor outcomes are insufficient. The purpose of this study is to assess the long term outcomes and risks that may arise from living kidney donation.

DETAILED DESCRIPTION:
Living donor transplants provide several advantages over deceased donor kidneys, including a shorter waiting time. Living donor grafts also appear to have a lower rate of delayed graft function and improved long-term recipient and graft survival. Most published studies of living kidney donation have supported that the donation process is relatively safe for the donor. However, these reports also emphasize concerns that comprehensive long-term data on U.S. live donor outcomes are insufficient. One concern is that current data may underestimate the true long-term morbidity and mortality of living kidney donation. Additionally, older studies might not apply to the current donor population that includes older and more obese individuals.

This is an observational study to look at the long term outcomes in living kidney donors. This study also seeks to find out if living kidney donors are at higher risk for certain conditions when compared to people of similar backgrounds who have not donated a kidney. Medical history, completed questionnaires, and blood and urine tests will be collected from donors and non donors. The compiled data from donors and non donors will be compared. Risks for diseases related to the kidney, heart, and blood vessels will be examined between the two groups. Quality of life and health insurance status will also be compared.

The study will be conducted in 2 phases. All donors who donated a kidney between 5 and 50 years ago at one of the three study transplant centers will be asked to take part in Phase 1. Phase 1 aims to collect limited medical information using a short questionnaire. Phase 2 will include Phase 1 donors who agree to further assessments and matched community control participants. Participants in Phase 2 will be asked to complete more in-depth questionnaires on health status and quality of life. Phase 2 also involves height, weight, and blood pressure measurements. Blood and urine will be collected for this study if the participant does not have the necessary tests within 3 years of study participation.

Seven thousand-eight hundred-sixty four (7864) previous kidney donors and about two thousand-five hundred (2500) control subjects will be asked to take part in this study. Participants will be recruited for this study over a 2.5.

ELIGIBILITY:
Inclusion Criteria:

* Underwent a unilateral donor nephrectomy between 5 and 50 years ago; but no later than June 30, 2005
* Alive at the time of study recruitment

Exclusion Criteria:

* Inability to contact donor

Community Control Inclusion Criteria:

* Matched to donor as healthy subject with a medical encounter date within 5 years of the date of donation and alive at the time of study recruitment
* Same gender as donor
* Same race as donor
* Matched by age, not to differ by more than 2 years
* Matched by BMI, not to differ by more than 5 kg/m^2 (JHS only)

Community Control Exclusion Criteria:

* Inability to contact control participant
* Inability or unwillingness to provide informed consent
* Hypertension or identified Charlson comorbidity index variable diagnosed prior to or on the encounter date matched to the donor date of donation (REP only)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants who have either donated a kidney or control subjects who are matched to have similar demographics and health condition a donor in the study.
Sampling Method: Non-Probability Sample
Enrollment: 7029 (Actual)
Dates: Start 2009-10; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Prevalence and incidence of hypertension, proteinuria, renal disease, and anemia | Since donation
Prevalence and incidence of cardiovascular disease as manifested by myocardial infarction (MI), heart failure (HF), stroke, and CABG/PTCA | Since donation
Quality of life and insurance status | Since donation

SECONDARY OUTCOMES:
Incidence of hypertension, proteinuria, renal disease, anemia, and QOL in black and white donors. | Since donation
Incidence of hypertension, proteinuria, renal disease, anemia, and QOL in donors with open nephrectomy and in donors with laparoscopic nephrectomy. | Since donation
The operative morbidity in living kidney donors with open nephrectomy and in donors with laparoscopic nephrectomy. | Since donation
Incidence of hypertension, proteinuria, renal disease, anemia, and QOL in standard living kidney donors and extended criteria donors. | Since donation
Incidence of hypertension, proteinuria, renal disease, anemia, and QOL in donors more than 20 years since donation and in donors between 5 and 20 years since donation. | Since donation
The identification of donor family characteristics that correlated with living kidney donor risk for morbidity and renal disease. | Retrospective
Donor physical health and recipient post-transplant course as it correlates with positive QOL scores and negative QOL scores. | Since donation
Identify the predictors and correlates of donors' quality of life outcomes | Throughout study
Compare post-donation blood pressures, estimated glomerular filtration rate (GFR), urine protein levels and hemoglobin levels with those derived from population-based studies and matched community control participants | After donation
Recipient outcomes for donors participating in the study and those who decline to participate. | After donation

CONTACTS AND LOCATIONS:
Overall Officials: Sandra J. Taler, MD, Principal Investigator — Mayo Clinic, Division of Nephrology and Hypertension
Locations (3):
- United States (3):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Bieniasz M, Domagala P, Kwiatkowski A, Gozdowska J, Krzysztof O, Kieszek RA, Trzebicki J, Durlik M, Rowinski W, Chmura A. The assessment of residual kidney function after living donor nephrectomy. Transplant Proc. 2009 Jan-Feb;41(1):91-2. doi: 10.1016/j.transproceed.2008.08.160. PMID 19249485
- [Background] Hernandez D, Alvarez A, Armas A, Rufino M, Porrini E, Torres A. [Metabolic syndrome and live kidney donor: is this syndrome a contraindication to donation?]. Nefrologia. 2009;29(1):20-9. doi: 10.3265/Nefrologia.2009.29.1.20.1.en.full.pdf. Spanish. PMID 19240768
- [Background] Horvat LD, Shariff SZ, Garg AX; Donor Nephrectomy Outcomes Research (DONOR) Network. Global trends in the rates of living kidney donation. Kidney Int. 2009 May;75(10):1088-98. doi: 10.1038/ki.2009.20. Epub 2009 Feb 18. PMID 19225540
- [Background] Rowinski W, Chmura A, Wlodarczyk Z, Ostrowski M, Rutkowski B, Domagala P, Dziewanowski K, Matych J, Durlik M, Grenda R. Are we taking proper care of living donors? A follow-up study of living kidney donors in Poland and further management proposal. Transplant Proc. 2009 Jan-Feb;41(1):79-81. doi: 10.1016/j.transproceed.2008.08.140. PMID 19249481
- [Result] Taler SJ, Messersmith EE, Leichtman AB, Gillespie BW, Kew CE, Stegall MD, Merion RM, Matas AJ, Ibrahim HN; RELIVE Study Group. Demographic, metabolic, and blood pressure characteristics of living kidney donors spanning five decades. Am J Transplant. 2013 Feb;13(2):390-8. doi: 10.1111/j.1600-6143.2012.04321.x. Epub 2012 Nov 8. PMID 23137211
- [Result] Jacobs CL, Gross CR, Messersmith EE, Hong BA, Gillespie BW, Hill-Callahan P, Taler SJ, Jowsey SG, Beebe TJ, Matas AJ, Odim J, Ibrahim HN; RELIVE Study Group. Emotional and Financial Experiences of Kidney Donors over the Past 50 Years: The RELIVE Study. Clin J Am Soc Nephrol. 2015 Dec 7;10(12):2221-31. doi: 10.2215/CJN.07120714. Epub 2015 Oct 13. PMID 26463883
- [Result] Jowsey SG, Jacobs C, Gross CR, Hong BA, Messersmith EE, Gillespie BW, Beebe TJ, Kew C, Matas A, Yusen RD, Hill-Callahan M, Odim J, Taler SJ; RELIVE Study Group. Emotional well-being of living kidney donors: findings from the RELIVE Study. Am J Transplant. 2014 Nov;14(11):2535-44. doi: 10.1111/ajt.12906. Epub 2014 Oct 7. PMID 25293374
- [Result] Gross CR, Messersmith EE, Hong BA, Jowsey SG, Jacobs C, Gillespie BW, Taler SJ, Matas AJ, Leichtman A, Merion RM, Ibrahim HN; RELIVE Study Group. Health-related quality of life in kidney donors from the last five decades: results from the RELIVE study. Am J Transplant. 2013 Nov;13(11):2924-34. doi: 10.1111/ajt.12434. Epub 2013 Sep 6. PMID 24011252
- [Result] Noppakun K, Cosio FG, Dean PG, Taler SJ, Wauters R, Grande JP. Living donor age and kidney transplant outcomes. Am J Transplant. 2011 Jun;11(6):1279-86. doi: 10.1111/j.1600-6143.2011.03552.x. Epub 2011 May 12. PMID 21564530
- [Result] Messersmith EE, Gross CR, Beil CA, Gillespie BW, Jacobs C, Taler SJ, Merion RM, Jowsey SG, Leichtman AB, Hong BA; RELIVE Study Group. Satisfaction With Life Among Living Kidney Donors: A RELIVE Study of Long-Term Donor Outcomes. Transplantation. 2014 Dec 27;98(12):1294-300. doi: 10.1097/TP.0000000000000360. PMID 25136843
- See also: National Institute of Allergy and Infectious Diseases (NIAID) website — https://www.niaid.nih.gov/
- See also: National Heart, Lung, and Blood Institute website — https://www.nhlbi.nih.gov/
- See also: National Kidney Registry website — http://www.kidneyregistry.org/
- Available data/document: Individual Participant Data Set: SDY290 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY290 — ImmPort study identifier is SDY290
- Available data/document: Study Protocol: SDY290 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY290 — ImmPort study identifier is SDY290
- Available data/document: Study summary, -design, -demographics, -files.: SDY290 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY290 — ImmPort study identifier is SDY290